CLINICAL TRIAL: NCT06792162
Title: Single Center, Phase II Clinical Study of PD-1 Antibody Carilizumab Combined with Apatinib for Unresectable Stage III and IV DMMR Gastric Cancer
Brief Title: PD-1 Antibody Carilizumab Combined with Apatinib for Unresectable Stage III and IV DMMR Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006761-M2022295
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib; spartalizumab

STUDY DESIGN:
Intervention Model Description: Drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PD-1 antibody Carilizumab combined with apatinib for unresectable dMMR gastric cancer (Experimental): Participants will receive Carilizumab 200mg repeated every 21 days and Apatinib 250mg everyday
  Interventions: Drug: Carilizumab and Apatinib

INTERVENTIONS:
Drug: Carilizumab and Apatinib — After every 2 cycles of meparticipants. Apatinib was discontinued for one cycle and an additional course of Carilizumab was administered in preparation for surgery. The time between the last dose and surgery was 3-6 weeks, with a maximum of 6 weeks. Both surgical and non-surgical participants will continue to receive treatment with the original regimen of Carilizumab combined with Apatinib after surgery until disease progression, recurrence, or death, for a maximum of 2 years.
  Other Names: PD-1 antibody

SUMMARY:
Evaluate the safety and efficacy of PD-1 antibody Carilizumab combined with apatinib for the conversion therapy of unresectable stage III and IV dMMR gastric cancer.

DETAILED DESCRIPTION:
This study is a prospective, open label, single center, phase II clinical trial aimed at evaluating the safety and efficacy of PD-1 antibody Carilizumab combined with apatinib for the conversion therapy of unresectable stage III and IV dMMR gastric cancer.

The study participants were unresectable stage III and IV dMMR gastric cancer patients who had not undergone any anti-tumor treatment. The study aims to enroll 20 participants with a primary endpoint of 1-year disease progression free survival rate. participants who meet the inclusion criteria will receive treatment with both Carilizumab and Apatinib, repeated every 21 days. During the conversion therapy period, the researchers evaluate whether surgery can be performed after every 2 cycles of medication for the subjects. After evaluation by the researchers, the participants were deemed eligible for surgery. Apatinib was discontinued for one cycle and an additional course of Carilizumab was administered in preparation for surgery. The time between the last dose and surgery was 3-6 weeks, with a maximum of 6 weeks. Both surgical and non-surgical subjects will continue to receive treatment with the original regimen of Carilizumab combined with Apatinib after surgery until disease progression, recurrence, or death, for a maximum of 2 years.

After the treatment is completed, a treatment end visit, a post treatment safety visit, and survival follow-up will be conducted. Participants who end the study due to non disease progression reasons will undergo imaging evaluation at the end of treatment (if no imaging evaluation has been received within 4 weeks before the end of treatment), and imaging evaluation will be conducted every 2 months after the end of treatment to assess the time of disease progression. After the completion of treatment, the participants will undergo a survival follow-up every 90 days to collect and record their survival status and subsequent anti-tumor treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years old, gender not limited;
2. Histologically confirmed unresectable stage III and IV dMMR (complete loss of at least one protein, MLH1, PMS2, MSH2, and MSH6), gastric adenocarcinoma (GC) (excluding neuroendocrine tumors) or gastroesophageal junction adenocarcinoma (GEJ);
3. Unresectable gastric cancer patients with potential for conversion therapy, defined as gastric cancer patients with single organ metastasis (such as liver metastasis, ovarian metastasis, lung metastasis), retroperitoneal lymph node metastasis, supraclavicular lymph node metastasis, localized peritoneal metastasis, invasion of surrounding organs, and other gastric cancer patients evaluated by researchers as feasible for conversion therapy;
4. Without surgery, radiation therapy, or immunotherapy for the gastric cancer lesion or metastatic tumor.
5. ECOG PS score 0-1 points;
6. Expected survival period ≥ 3 months;
7. The main organ functions are normal, and there are no severe abnormalities in blood, heart, lung, liver, kidney, bone marrow, or immunodeficiency diseases.
8. Normal coagulation function, no active bleeding or thrombotic diseases:
9. The time from the end of traditional Chinese medicine, traditional Chinese patent medicines and simple preparations and immunomodulator (such as thymosin, interleukin, etc.) that have used anti-tumor drugs in the past to the start of the study must be ≥ 2 weeks;
10. Non surgical sterilization or female subjects of childbearing age are required to use a medically approved contraceptive measure (such as intrauterine device, contraceptive pill, or condom) during the study treatment period and within 180 days after the end of the study treatment; Female subjects of childbearing age who undergo non-surgical sterilization must have a negative serum HCG test within 72 hours prior to randomization; And it must be during non lactation period; For male participants whose partners are women of childbearing age, effective contraception methods should be used during the study treatment period and within 180 days after the end of the study treatment period.
11. Subjects voluntarily participated in this study, fully understood and informed of the study, and signed the Informed Consent Form (ICF);

Exclusion Criteria:

1. Other malignant tumors have been diagnosed within 5 years before the first use of the investigational drug, except for effectively treated skin basal cell carcinoma, skin squamous cell carcinoma and/or effectively resected cervical carcinoma in situ and/or breast cancer and/or thyroid cancer and other malignant tumors that have achieved long-term survival;
2. Suffering from any active autoimmune disease or history of autoimmune disease, such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (except for patients with stable hormone levels after treatment); Subjects with childhood asthma who have been completely relieved and do not require any intervention or vitiligo in adulthood may be included, but those who require medical intervention with bronchodilators may not be included;
3. People with congenital or acquired immune deficiency, such as people infected with human immunodeficiency virus (HIV), active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody is positive, and HCV-RNA is higher than the detection limit of the analytical method) or people with co infection of hepatitis B and hepatitis C;
4. Within 14 days prior to the first use of the investigational drug, immunosuppressive drugs have been used, excluding nasal and inhaled corticosteroids or systemic corticosteroids at physiological doses (i.e. not exceeding 10 mg/day of prednisolone or other corticosteroids at physiological doses of equivalent drugs);
5. Vaccination with attenuated live vaccine within 4 weeks before the first administration or planned during the study period;
6. Patients with hypertension who cannot be reduced to normal range by antihypertensive medication (systolic blood pressure ≤ 140 mmHg/diastolic blood pressure ≤ 90 mmHg);
7. Suffering from uncontrolled clinical symptoms or diseases of the heart, such as (1) NYHA class II or above heart failure, (2) unstable angina, (3) myocardial infarction within 1 year, (4) poorly controlled arrhythmia;
8. Patients who have had or currently have interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, etc., and whose lung function is severely impaired, which may interfere with the detection and management of suspected drug-related pulmonary toxicity;
9. suffer from active pulmonary tuberculosis;
10. Severe infection (such as requiring intravenous infusion of antibiotics, antifungal or antiviral drugs) within 4 weeks before the first medication, or unexplained fever (body temperature ≥ 38.5 ° C) during the screening period/before the first administration;
11. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
12. Those who are known to have a history of allergies to the components of this drug regimen;
13. There is a possibility of increasing participation in research and medication risks, or other severe, acute, and chronic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
The rate of 1-year PFS | From enrollment to the end of treatment at 1year"
  The progression free survival (PFS) was defined as the time from the beginning of systematic anti-cancer therapy to disease progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Baoshan Cao, Principal Investigator — Department of Medical Oncology and Radiation Sickness, Peking University Third Hospital
Locations (1):
- Peking University third hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The datasets analyzed during the study are available on reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the trial is completed
Access Criteria: Used for scientific research